CLINICAL TRIAL: NCT02865122
Title: A Multi-Center, Randomized, Double-Blind, Three-Arm, Parallel-Group Trial to Assess the Efficacy and Safety of NTRA-9620 in Infants With Short Bowel Syndrome (SBS) Following Surgical Resection
Brief Title: Safety and Efficacy Study in Infant With SBS
Acronym: GIFT
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Sponsor decision based on enrollment
Sponsor: Elgan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GIFT-02
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- NTRA-9620-A (Experimental): NTRA-9620 Dose 1 To be dosed orally for 24 weeks, 4 times/day
  Interventions: Drug: NTRA-9620
- NTRA-9620-B (Experimental): NTRA-9620 Dose 2 To be dosed orally for 24 weeks, 4 times/day
  Interventions: Drug: NTRA-9620
- Placebo (Placebo Comparator): Placebo To be dosed orally for 24 weeks, 4 times/day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NTRA-9620 — Oral daily dose
  Arms: NTRA-9620-A; NTRA-9620-B
Drug: Placebo — Oral daily dose
  Arms: Placebo

SUMMARY:
The objective of this clinical study is to evaluate the efficacy and safety of NTRA-9620 compared with placebo in pediatric subjects (aged 28 weeks postmenstrual age to 52 weeks old) with SBS following surgical resection

ELIGIBILITY:
Inclusion Criteria

1. Subject must be at least 28 weeks post-menstrual age and up to 52 weeks chronological age at enrollment.
2. Subject weight must be at least 500 grams (17.6 ounces) at time of enrollment.
3. After major surgical resection leading to SBS, the subject has maximally 70% of expected bowel length preserved or an ostomy in place such that ≤ 70% of the small bowel is available for nutrient absorption.

Exclusion Criteria

1. Subject has undergone any bowel lengthening procedure.
2. Subject has a malabsorption disorder due to:

   * congenital etiology (such as microvilli inclusion disease, tufting enteropathy)
   * Untreated Hirchsprung's disease
3. Uncontrolled systemic infection, acute gastroenteritis, pneumonia, cardiovascular or other abnormality including EKG findings that in the opinion of the investigator makes the infant unstable and at significant risk of not completing first 12 weeks of the study.
4. Subjects with hyperinsulinemia.
5. Subjects with unexplained or recurrent hypoglycemia with blood glucose ≤ 50 mg/dL within 48 hours of treatment initiation.

Ages: 2 Weeks to 52 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-03-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Lucile Packard Children's Hospital Stanford, Palo Alto, California
  - Connecticut Children's Hospital, Hartford, Connecticut
  - University of Florida, Gainesville, Florida
  - Children's Mercy Hospital, Kansas City, Missouri
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Texas Children's Hospital, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- NTRA-9620-A: NTRA-9620 Dose 1: 2 IU/kg To be dosed orally for 24 weeks, 4 times/day
  NTRA-9620: Oral daily dose
- NTRA-9620-B: NTRA-9620 Dose 2 - 1 IU/kg To be dosed orally for 24 weeks, 4 times/day
  NTRA-9620: Oral daily dose
Period: Overall Study
Arm/Group | NTRA-9620-A | NTRA-9620-B | Placebo
Started | 1 | 1 | 0
Completed | 0 | 1 | 0
Not Completed | 1 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects randomized to placebo. Study was terminated early.
Groups:
- Total: Total of all reporting groups
Arm/Group | NTRA-9620-A | NTRA-9620-B | Placebo | Total
Number analyzed (Participants) | 1 | 1 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 1 |  | 2
  Between 18 and 65 years | 0 | 0 |  | 0
  >=65 years | 0 | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 1 | 1 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 1 | 0 |  | 1
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in %PN/IV
Description: Percent change in %PN/IV from baseline based on caloric intake
Time Frame: baseline and end of treatment or 24 weeks, whichever occurs first
Population: During the course of the study only two (2) subjects were enrolled prior to discontinuation. Thus, no conclusions regarding the efficacy or safety (risk/benefit) of NTRA-9620 in the short bowel syndrome (SBS) population can be determined from this study.
Arm/Group | NTRA-9620-A | NTRA-9620-B | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Only one patient experienced Serious Adverse Events. There were no deaths in the study. There were no "Other" Adverse Events experienced in the study.
Arm/Group | NTRA-9620-A | NTRA-9620-B | Placebo
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NTRA-9620-A (N=1) | NTRA-9620-B (N=1) | Placebo (N=0)
Apparent life threatening event (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 0 (0) | 0 (0) — Aspiration Neonatal respiratory distress system Pulmonary hypertension Pulmonary vein stenosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-10): https://cdn.clinicaltrials.gov/large-docs/22/NCT02865122/Prot_SAP_001.pdf